CLINICAL TRIAL: NCT01199419
Title: Cost-effectiveness of Percutaneous Coronary Intervention With TAXUS Stents in Patients With Multivessel Coronary Artery Disease Compared With Aortocoronary Bypass Surgery 5 Years After Intervention
Brief Title: Cost-effectiveness of PCI With Taxus vs CABG - 5 Years FUP
Status: Completed | Type: Observational
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Mariann Gyongyosi, MD PhD, Medical University of Vienna
Other Study IDs: Version 1
Record Dates: First submitted 2010-09-09; First posted 2010-09-13 (Estimated); Last update posted 2014-07-18 (Estimated); Status verified 2014-07

CONDITIONS: Multivessel Coronary Artery Disease
Keywords: multivessel coronary artery disease; drug-eluting stent; CABG; cost-effectiveness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (2):
- PCI
  Interventions: Procedure: comparison of PCI vs. CABG in multivessel disease
- CABG
  Interventions: Procedure: comparison of PCI vs. CABG in multivessel disease

INTERVENTIONS:
Procedure: comparison of PCI vs. CABG in multivessel disease — invasive treatment of coronary artery disease

SUMMARY:
The objective of the present study is to analyze the cost-effectiveness of percutaneous coronary intervention (PCI) using TAXUS stents compared to the costs of coronary artery bypass surgery (CABG) in patients with multivessel coronary artery disease (CAD) in the first 5 years and then 10 years after intervention. Multivessel PCI or CABG was performed in 114 or 93 patients, respectively. Clinical outcomes, in terms of incidence of acute myocardial infarction (AMI), all-cause death, target vessel revascularization (TVR) and stroke, resource use and costs are analyzed prospectively over a 5 and 10-year follow-up (FUP) period. Overall costs consist of the baseline costs of the index procedure (PCI or CABG), clinical and angiographic procedure-related treatments during the entire FUP. The primary endpoint is cost-effectiveness and clinical effectiveness, defined as the reduction of the composite of major adverse cardiac and cerebrovascular events (MACCE).

ELIGIBILITY:
Inclusion Criteria:

* two or three-vessel disease requiring percutaneous or surgical multivessel intervention with the aim of complete revascularization
* age > 18 years
* clinical symptoms (stable or unstable angina) or signs of myocardial ischemia
* ≥ 50% diameter stenosis of each lesion

Exclusion Criteria:

* acute myocardial infarction (< 48 h);
* contraindications to clopidogrel, aspirin, heparin and taxol;
* pregnancy or lack of protection against pregnancy or breast-feeding during the study;
* hemorrhagic diathesis and platelet count <100.000/ml3

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients, treated with multivessel disease requiring revascularization were consecutively included in this study.
Sampling Method: Probability Sample
Enrollment: 207 (Actual)
Dates: Start 2004-01; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Cost-effectiveness of percutaneous coronary intervention with Taxus stents compared to CABG in patients with multivessel coronary artery disease. | in-hospital phase (up to 3 weeks)
Cost-effectiveness of percutaneous coronary intervention with Taxus stents compared to CABG in patients with multivessel coronary artery disease. | 6 months
Cost-effectiveness of percutaneous coronary intervention with Taxus stents compared to CABG in patients with multivessel coronary artery disease. | 12 months
Cost-effectiveness of percutaneous coronary intervention with Taxus stents compared to CABG in patients with multivessel coronary artery disease. | 5 years
Cost-effectiveness of percutaneous coronary intervention with Taxus stents compared to CABG in patients with multivessel coronary artery disease. | 10 years

SECONDARY OUTCOMES:
Occurrence of MACCE, defined as cardiac death, nonfatal myocardial infarction, target vessel revascularization and stroke | 6 months
Rate of target vessel revascularization | 6 months
Occurrence of non-fatal acute myocardial infarction | 6 months
Occurrence of cardiac death | 6 months
Calculation of the total costs | in-hospital phase (up to 3 weeks)
Occurrence of MACCE, defined as cardiac death, nonfatal myocardial infarction, target vessel revascularization and stroke | 12 months
Occurrence of MACCE, defined as cardiac death, nonfatal myocardial infarction, target vessel revascularization and stroke | 5 years
Occurrence of MACCE, defined as cardiac death, nonfatal myocardial infarction, target vessel revascularization and stroke | 10 years
Rate of target vessel revascularization | 12 months
Rate of target vessel revascularization | 5 years
Rate of target vessel revascularization | 10 years
Occurrence of non-fatal acute myocardial infarction | 12 months
Occurrence of non-fatal acute myocardial infarction | 5 years
Occurrence of non-fatal acute myocardial infarction | 10 years
Occurrence of cardiac death | 12 months
Occurrence of cardiac death | 5 years
Occurrence of cardiac death | 10 years
Calculation of the total costs | 6 months
Calculation of the total costs | 12 months
Calculation of the total costs | 5 years
Calculation of the total costs | 10 years

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of Vienna, Dept. of Cardiology, Vienna, Austria